CLINICAL TRIAL: NCT04417140
Title: A Prospective, Double-Blinded, Randomized Controlled Trial of Dehydrated Human Amniotic-Chorionic Membrane for Incisional Hernia Prophylaxis
Brief Title: A Prospective, Double-Blinded, Randomized Controlled Trial of dHACM for Incisional Hernia Prophylaxis
Acronym: NO-HERNIA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Collaborators: LSUHSC-NO (Unknown)
Responsible Party: Principal Investigator, Frank Lau, MD, Associate Professor of Plastic & Reconstructive Surgery, Louisiana State University Health Sciences Center in New Orleans
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LSUHSC-NO IRB # 19-174
Record Dates: First submitted 2020-06-02; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Incisional Hernia
Keywords: amniotic membrane; placenta-derived tissue; incisional hernia
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Intervention Model Description: 5.1 General Design Description A double-blinded RCT with two arms: treatment (dHACM) and control. Patients will be recruited from LSUHSC-NO surgeons' practices .
  Subjects will be randomized to treatment or control at a rate of 1:1, stratified by surgeon. Subjects, nursing staff, and surgeons not present at the time of fascial closure will be kept blinded to the subjects' treatment arm. Computer-generated randomization will be performed in permutated blocks of 20 patients, using SAS version 9.4.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: 5.1 General Design Description A double-blinded RCT with two arms: treatment (dHACM) and control. Patients will be recruited from 8 LSUHSC-NO surgeons' practices (Drs. Boudreaux, Stuke, Orangio, Moore, tMarr, Hunt, Greiffenstein, and Barton).
  Subjects will be randomized to treatment or control at a rate of 1:1, stratified by surgeon. Subjects, nursing staff, and surgeons not present at the time of fascial closure will be kept blinded to the subjects' treatment arm. Computer-generated randomization will be performed in permutated blocks of 20 patients, using SAS version 9.4.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Arm-dHACM (Experimental): Patients enrolled in this arm will have a thin sheet of dHACM placed as an overlay over the length of the closed incisions. dHACM is Dehydrated Human Amniotic-Chorion Membrane. It is a FDA registered healing adjunct that has been applied in a broad range of diseases including wounds, plantar fasciitis and burns.
  Interventions: Biological: dHACM (AmnioWrap)
- Control Arm (No Intervention): Patients enrolled in this arm will have routine closure.

INTERVENTIONS:
Biological: dHACM (AmnioWrap) — Dehydrated human amnion-chorion membrane (dHACM) is a healing adjunct that has been applied in a broad range of disease, and is FDA registered for wound healing.
  Arms: Treatment Arm-dHACM

SUMMARY:
Currently, no standard of care exists to prevent incisional hernias (IH). This study will compare how frequently IH develop in standard abdominal closures vs. abdominal closures with dHACM added. By adding dHACM to the standard closure, we think we can reduce the formation of IH.

If patients decide to participate in this study, they will be randomly assigned to one of two study arms, Arm A or Arm B. They will have a 50% chance of being assigned to either arm. The assignment will be made by computer program and is completely random. Patients are not informed of which arm they are assigned.

Arm A (Treatment Arm): dHACM Patients enrolled in this arm will have a thin sheet of dHACM placed as an overlay over the length of the closed incisions. dHACM is Dehydrated Human Amniotic-Chorion Membrane. It is a FDA-registered healing adjunct that has been applied in a broad range of diseases including wounds, plantar fasciitis and burns.

Arm B (Control Arm) Patients enrolled in this arm will have standard fascial closure.

Data collection will be performed at routine follow-up outpatient clinic visits with the primary surgeon to assess for IH related symptoms. At 6 months after surgery, patients will see a surgeon who is blinded to the randomization. This surgeon will perform a painless handheld ultrasound examination of the incision site.

DETAILED DESCRIPTION:
Two million laparotomies are performed annually in the United States (US). Following these surgeries, the incidence of new incisional hernias (IH) is estimated at 400,000 cases per year. These hernias are a major source of morbidity and mortality for patients, and they result in $6-10 billion per year in healthcare costs. Our multidisciplinary hernia prevention group has identified a novel IH prevention strategy in the form of dehydrated human amniotic-chorionic membrane (dHACM). We previously showed that dHACM prevents IH in animal models, and subsequently in a prospective cohort of high-risk patients.

The purpose of this trial is to quantify the efficacy of dHACM in IH prophylaxis by performing a prospective, double-blinded randomized controlled trial. Our specific aim is to test the hypothesis that augmentation of standard abdominal fascia closures with prophylactic, onlay dHACM sheets without fixation will reduce IH formation in a high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 years
* Written informed consent
* Non-emergent operation
* Predicted incisional herna (IH) risk ≥150% of the average IH risk, as calculated by the University of Pennsylvania Hernia Risk Calculator, which accounts for 18 IH risk factors
* BMI > 27 yields IH risk > 150% of the average IH risk; this can be used as a shortcut for screening potential subjects

Exclusion Criteria:

* Previous intraperitoneal mesh placement
* Previous abdominal incisional hernia
* Emergency procedures
* Patients with inflammatory bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 533 (Estimated)
Dates: Start 2020-05-20 (Actual); Primary Completion 2022-05-20 (Estimated); Study Completion 2022-05-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of IH as determined by physical exam or abdominal ultrasound demonstrating a midline fascial defect and hernia sac> 4mm diameter | 6 months

SECONDARY OUTCOMES:
Intraoperative and postoperative complications | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No